CLINICAL TRIAL: NCT06747689
Title: Effect of Sleep Quality on Self-Care in Patients with Heart Failure: a Longitudinal Analysis
Brief Title: Association Between Sleep Quality and Self-Care in Heart Failure Patients
Status: Recruiting | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Arzu AKBABA, Principal Investigator, Dokuz Eylul University
Other Study IDs: 2024/41-11
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure; Sleep Quality; Self Care; Cognitive Function
MeSH Terms: conditions — Heart Failure; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The research will be conducted as a prospective and relational study to longitudinally investigate the effect of sleep quality on self-care in patients with heart failure (HF) and to evaluate the relationship between self-care, sleep quality, and cognitive functions. The sample size was calculated using the multiple linear regression model with the G*Power Version 3.1 program. Based on a medium effect size of 0.15, an alpha of 0.05, a power of 0.95, and 18 predictors, the sample size was determined to be 188. Considering a potential dropout rate of 10%, it was decided to complete the study with a minimum of 207 participants.

Data will be collected from patients who apply to the Dokuz Eylül University Cardiology Outpatient Clinic and meet the inclusion criteria. After signing the informed consent form, participants will be followed up at baseline, the 1st month, the 3rd month, and the 6th month by telephone. The Statistical Package for Social Sciences (SPSS) 24.0 will be used to analyze the numerical data of the research. Descriptive statistics, including number, percentage, mean, and standard deviation, as well as inferential statistics such as the χ2 test, t-test for independent groups, and multiple linear regression, will be employed in the data analysis.

ELIGIBILITY:
The study will include patients who:

* Are diagnosed with heart failure according to international guidelines,
* Are aged 18 years or older,
* Can communicate via phone, and
* Are willing to participate in the study.

Exclusion Criteria:

The study will exclude patients who:

* Have been hospitalized within one month prior to inclusion,
* Have experienced major psychological trauma or stress in the last three months,
* Have serious comorbidities or malignant cancers,
* Have advanced hearing impairment,
* Are using prescription drugs for insomnia or psychiatric conditions,
* Work night shifts, or
* Reside in nursing homes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the cardiology clinic of Dokuz Eylül University Hospital.
Sampling Method: Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | From December 2024 to January 2026
  The Pittsburgh Sleep Quality Index (PSQI) was developed by Buysse and colleagues in 1989. It is a scale that provides a quantitative measurement of sleep quality, distinguishing between good and poor sleep. Its validity and reliability study was conducted in Turkey in 1996 by Agargün and colleagues, with a Cronbach's alpha value of.80. The scale is a four-point Likert type and contains a total of 24 questions, comprising seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. Each component is scored between 0 and 3 based on the frequency of symptoms. The sum of the seven component scores yields the total PSQI score, which ranges from 0 to 21. A total score of 5 or above indicates poor sleep quality and a high level of sleep disturbance.
Self Care | From December 2024 to January 2026
  Self-care will be assessed using the nine-item version of the European Heart Failure Self-Care Behavior Scale (Jaarsma et al., 2003). The validity and reliability of the scale in our country were established by Yıldız and Erci (Yıldız & Erci, 2018). This Likert-type scale measures self-care behaviors such as recognizing symptoms like edema, dyspnea, and fatigue related to HF, adhering to regular medication use, monitoring weight, and restricting fluid and salt intake. Participants are asked to choose one of the following options for each item: completely agree (1), agree (2), undecided (3), disagree (4), or completely disagree (5). A higher total score indicates lower self-care, while a lower score indicates higher self-care. Fit measures for the Structural Equation Model of the scale include RMSEA = 0.047 (CI = 0.00-0.079), AGFI = 0.83, and GFI = 0.91 (Jaarsma et al., 2003). In the study by Yıldız and Erci, the Cronbach's alpha coefficient was reported as 0.82 (Yıldız & Erci,2018)

SECONDARY OUTCOMES:
Cognitive Fuction | From December 2024 to January 2026
  The Telephone Cognitive Screening Test (T-KogS) was adapted from the ALFI-Mini Mental Assessment test by Newkirk and colleagues. This scale can be administered face-to-face to assess the cognitive functions of Alzheimer's patients or used in situations where face-to-face interviews are not possible (Newkirk et al., 2004). The T-KogS evaluates cognitive domains including orientation (e.g., year, season, day, day of the week, month, state, county, city/town, address, and telephone number), registration and recall (e.g., recalling three objects: apple, table, penny), attention (e.g., writing the word "WORLD" backwards), and language (e.g., repetition of "no if, and, or but," single object naming, and a three-step command). The total score on the T-KogS ranges from 0 to 26, with higher scores indicating better cognitive performance. The Turkish validity and reliability study of the scale was conducted by Naharci et al. in 2020, and the Cronbach's alpha value was reported as 0.73.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No